CLINICAL TRIAL: NCT02273661
Title: Evaluation of a Therapeutic Strategy Including Nebulised Liposomal Amphotericin B (Ambisome®) in Maintenance Treatment of Allergic Bronchopulmonary Aspergillosis (Cystic Fibrosis Excluded)
Acronym: NEBULAMB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEBULAMB
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Placebo Comparator): An aerosol of isotonic saline x 1/ week will be administered during 6 months
  Interventions: Drug: placebo
- Ambisome (Experimental): An aerosol of Liposomal Amphotericin B (Ambisome®) at 25 mg x 1/ week will be administered during 6 months
  Interventions: Drug: Liposomal amphotericin B (Ambisome®)

INTERVENTIONS:
Drug: Liposomal amphotericin B (Ambisome®) — An aerosol of Liposomal Amphotericin B (Ambisome®) at 25 mg x 1/ week will be administered during 6 months
  Arms: Ambisome
Drug: placebo — An aerosol of isotonic saline x 1/ week will be administered during 6 months
  Arms: Control

SUMMARY:
Compare the incidence of severe clinical exacerbations in the treatment of ABPA, between a strategy with a maintenance treatment and a conventional strategy without antifungal maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

All patients with ABPA justifying an attack treatment with corticosteroids and itraconazole and combining the following criteria:

1. atopic subject or a history of asthma , history of total Immunoglobin E (IgE)> 417 kU / L (or > 210 kU / L with a clear worsening) of a known ABPA), specific Immunoglobin E against Aspergillus fumigatus positive ( >0.35 KUA/L) or positive skin tests.
2. associated with two other of the following criteria: documentation of precipitating antibodies or Immunoglobulin G positive to Aspergillus fumigatus, of radiological infiltrates associated with ABPA (transitional / persistent / bronchial dilation), of blood eosinophilia > 500 elements/mm3.
3. After informing and obtaining consent signed.

Exclusion Criteria:

* Women of childbearing age who do not have an effective contraception for at least 12 first months of the study( 10 months + 2 months of treatment washout) pregnant or lactating women,
* Patient with cystic fibrosis
* Patient with a contra-indication to itraconazole
* Intolerance to β2 -agonists
* Known hypersensitivity to liposomal amphotericin B or any other component
* Laboratory abnormalities: significant abnormalities of platelet blood count , liver function tests (SGPT, SGOT(serum glutamate oxaloacetate transaminase) , total bilirubin > 5 times the upper limit of the normal range )
* severe renal function impairment (creatinine clearance enf to 30 ml/min)
* Concomitant use of one or more of the following treatments: Alfuzosine, alcaloïdes de l'ergot de seigle vasoconstricteur, aliskiren, astemizole, atorvastatine, avanafil, association Ombitasvir and Paritaprevir, Bepridil, Cisaprid, Dabigatran, dapoxetin, domperidon, dronedaron, Eplerenone, Halofantrin, Ivabradin, Lomitapid, lurasidon, Millepertuis, mizolastin, Pimozid,Quétiapin, quinidin, Ranolazine, ritonavir, Sertindole, sildénafil, simvastatin, sirolimus, Sultoprid, Terfenadine, ticagrelor, triazolam Vardénafil (in men over than 75)
* patient with anti IgE- monoclonal antibody for less than 4 months or with current complications related to previous treatment with anti IgE- monoclonal antibody -
* Ventricular dysfunction demonstrated such as congestive heart failure or a history of congestive heart failure
* Simple aspergilloma, chronic pulmonary aspergillosis, invasive pulmonary aspergillosis
* Respiratory infection aggravating asthma or ABPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
occurrence of first severe clinical exacerbation | within 24 months following the attack treatment,
  Occurrence of severe clinical exacerbation within 24 months following attack treatment, defined by the onset or worsening of dyspnea aggravating the baseline condition that justified:
  1. -increased inhalation treatments (inhaled bronchodilators and / or corticosteroids)
     * and / or initiation of systemic corticosteroid treatment
     * and / or hospitalization
  2. AND persisting for more than 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France

REFERENCES:
- [Derived] Godet C, Brun AL, Couturaud F, Laurent F, Frat JP, Marchand-Adam S, Gagnadoux F, Blanchard E, Taille C, Philippe B, Hirschi S, Andrejak C, Bourdin A, Chenivesse C, Dominique S, Mangiapan G, Murris-Espin M, Riviere F, Garcia G, Blanc FX, Goupil F, Bergeron A, Flament T, Priou P, Mal H, de Keizer J, Ragot S, Cadranel J; NebuLamB Study Group and GREPI Network. CT Imaging Assessment of Response to Treatment in Allergic Bronchopulmonary Aspergillosis in Adults With Bronchial Asthma. Chest. 2024 Jun;165(6):1307-1318. doi: 10.1016/j.chest.2024.02.026. Epub 2024 Feb 20. PMID 38387646
- [Derived] Godet C, Couturaud F, Marchand-Adam S, Pison C, Gagnadoux F, Blanchard E, Taille C, Philippe B, Hirschi S, Andrejak C, Bourdin A, Chenivesse C, Dominique S, Bassinet L, Murris-Espin M, Riviere F, Garcia G, Caillaud D, Blanc FX, Goupil F, Bergeron A, Gondouin A, Frat JP, Flament T, Camara B, Priou P, Brun AL, Laurent F, Ragot S, Cadranel J; NebuLamB study group and GREPI network; Godet C, Couturaud F, Cadranel J, Frat JP, Brun AL, Laurent F, Marchand-Adam S, Pison C, Gagnadoux F, Blanchard E, Taille C, Philippe B, Hirschi S, Andrejak C, Chenivesse C, Dominique S, Bassinet L, Murris-Espin M, Riviere F, Garcia G, Caillaud D, Blanc FX, Goupil F, Gondouin A, Flament T, Camara B, Priou P, Ragot S. Nebulised liposomal amphotericin-B as maintenance therapy in allergic bronchopulmonary aspergillosis: a randomised, multicentre trial. Eur Respir J. 2022 Jun 16;59(6):2102218. doi: 10.1183/13993003.02218-2021. Print 2022 Jun. PMID 34764182